CLINICAL TRIAL: NCT03878485
Title: Pilot Study of Same-session MR-only Simulation and Treatment With Stereotactic MRI-guided Adaptive Radiotherapy (SMART) for Oligometastases of the Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201903023
Record Dates: First submitted 2019-03-14; First posted 2019-03-18 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Oligometastases of the Spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stereotactic MRI-guided Adaptive Radiotherapy (Experimental): -Radiotherapy will consist of stereotactic body therapy to the spine, to be given over either a two or five fraction course, delivered once daily or once every other day for a period of one to two weeks, for a total of two or five treatments (depending on whether a 2 or 5 fraction course is selected).
  Interventions: Device: MRIdian Linac System from ViewRay; Radiation: Stereotactic MRI-guided Adaptive Radiotherapy

INTERVENTIONS:
Device: MRIdian Linac System from ViewRay — * 0.35T MRI combined with a linear accelerator
  * This device will be used for the Stereotactic MRI-guided Adaptive Radiotherapy
  Other Names: MR-linac
Radiation: Stereotactic MRI-guided Adaptive Radiotherapy — -The MR-linac will be delivering the radiation
  Other Names: SMART

SUMMARY:
In light of the increasing experience with magnetic resonance image-guided radiotherapy (MRgRT) and adaptive planning and advances in magnetic resonance (MR)-only planning, the investigators propose here to evaluate the feasibility and safety of same-session MR-only simulation and treatment with SMART for spinal metastases. Although spine SBRT is a standard-of-care treatment modality, this expedited same-session MR-only simulation and treatment with SMART workflow is novel. Previously, delivery of spine SBRT has typically required several days from time of consultation to simulation and then 1-2 weeks from simulation to the initiation of treatment. On this proposed study, patients will not undergo computed tomography (CT) simulation and will instead have same-session MR-only simulation and treatment planning, on-table, using SMART. In this manner, patients would initiate treatment within just several days from the consult. Feasibility of the workflow will be defined as successful delivery of the first fraction of same-session MRI-only simulation and treatment with SMART on the first on-table attempt for at least 70% of patients. Patients will be treated in five fractions over 1-2 weeks. Although the long-term goal will be to achieve a significantly shortened time from consult to treatment as compared to traditional stereotactic body radiation therapy (SBRT) using simulation, the present study will be driven by short-term goals of workflow feasibility and safety.

ELIGIBILITY:
Inclusion Criteria:

* At least one disease site deemed to be suitable for treatment with spine SBRT as per radiation oncology evaluation.
* Karnofsky Performance Status (KPS) ≥ 60.
* Deemed medically fit for SBRT by treating physician
* Diagnostic CT with images through the projected treatment area within six months prior to enrollment.
* At least 18 years of age.
* Ability to understand and willingness to sign an IRB approved written informed

Exclusion Criteria:

* Past history of radiotherapy within the projected treatment field to be treated by MRI-guided SBRT
* Medical contraindication to undergoing MR imaging.
* Spine metastasis resulting in symptomatic spinal cord compression.
* Any other condition that, in the opinion of the treating radiation oncologist, renders the patient unfit for SBRT.
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-11-06 (Actual); Primary Completion 2023-10-09 (Actual); Study Completion 2024-01-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clifford Robinson, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stereotactic MRI-guided Adaptive Radiotherapy
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic MRI-guided Adaptive Radiotherapy
Number analyzed (Participants) | 10
Age, Continuous [Median (Full Range); unit: years] | 63 [26 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 10
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants to Receive Delivery of the First Fraction of Same-session MRI-only Simulation and Treatment With SMART on the First On-table Attempt
Time Frame: First on-table attempt of first fraction of radiation (an average of 1 day)
Measure: Count of Participants; unit: Participants
Arm/Group | Stereotactic MRI-guided Adaptive Radiotherapy
Number analyzed (Participants) | 10
Participants | 8

ADVERSE EVENTS:
Time Frame: Adverse events and all-cause mortality were collected from start of treatment through 3-month post-treatment follow-up visit.
Description: The following adverse events were not collected: grade 1-2 events regardless of relatedness, grade 3-4 events that predate SBRT, and grade 3-4 events that are not at least probably attributable to treatment.
Arm/Group | Stereotactic MRI-guided Adaptive Radiotherapy
All-Cause Mortality (participants affected / at risk) | 1/10
Serious Adverse Events (participants affected / at risk) | 2/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic MRI-guided Adaptive Radiotherapy (N=10)
Back pain (Musculoskeletal and connective tissue disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Stereotactic MRI-guided Adaptive Radiotherapy (N=10)
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-02-27): https://cdn.clinicaltrials.gov/large-docs/85/NCT03878485/Prot_SAP_000.pdf